CLINICAL TRIAL: NCT07314021
Title: Comparison of the Structured FEMOB Mobilization Technique and the MOPEXE Exercise Model in Women With Primary Dysmenorrhea
Brief Title: Primary Dysmenorrhea and Mobilization.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, ZEYNEP BETÜL BİLGİ, physiotherapist, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-4605
Record Dates: First submitted 2025-12-04; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Primary Dysmenorrhea
Keywords: mobilization; primary dysmenorrhea; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FEMOB (Active Comparator): Transcutaneous Electrical Nerve Stimulation (TENS) treatment will be applied to the lumbar and suprapubic areas using 2 channels and 4 electrodes. Conventional TENS (120 Hz) will be applied simultaneously to the lumbar and suprapubic areas for 30 minutes. Hot pack application will be done sequentially to the lumbar and suprapubic areas for 15 minutes each, for a total of 30 minutes.
  FEMOB is a mobilization model that includes temporo-mandibular, occipito-sacral, and sacroiliac joint mobilizations along with abdominal myofascial release and kinesio taping.
  Interventions: Other: MOPEXE; Other: CONTROL
- MOPEXE (Active Comparator): Transcutaneous Electrical Nerve Stimulation (TENS) treatment will be applied to the lumbar and suprapubic areas using 2 channels and 4 electrodes. Conventional TENS (120 Hz) will be applied simultaneously to the lumbar and suprapubic areas for 30 minutes. Hot pack application will be done sequentially to the lumbar and suprapubic areas for 15 minutes each, for a total of 30 minutes.
  5 minute-Meditation Therapy 10 minute-Progressive Relaxation training ( Bernstein-Borkovec Method) 5 min - Breathing Exercises (Diaphragmatic Breathing Exercise, Pursed lip breathing Exercise) 35 min -Motor Imagery Technique Focused Pelvic Floor Exercises-MOPEXE 5 min - Meditation Therapy Twice a week for 60 minutes 12 weeks Participants will be evaluated online at the beginning of the research and at the end of the 12-week program.
  Interventions: Other: FEMOB; Other: CONTROL
- CONTROL (Other): Transcutaneous Electrical Nerve Stimulation (TENS) treatment will be applied to the lumbar and suprapubic areas using 2 channels and 4 electrodes. Conventional TENS (120 Hz) will be applied simultaneously to the lumbar and suprapubic areas for 30 minutes. Hot pack application will be done sequentially to the lumbar and suprapubic areas for 15 minutes each, for a total of 30 minutes.
  Interventions: Other: FEMOB; Other: MOPEXE

INTERVENTIONS:
Other: FEMOB — Transcutaneous Electrical Nerve Stimulation (TENS) treatment will be applied to the lumbar and suprapubic areas using 2 channels and 4 electrodes. Conventional TENS (120 Hz) will be applied simultaneously to the lumbar and suprapubic areas for 30 minutes. Hot pack application will be done sequentially to the lumbar and suprapubic areas for 15 minutes each, for a total of 30 minutes. FEMOB is a mobilization model that includes temporo-mandibular, occipito-sacral, and sacroiliac joint mobilizations along with abdominal myofascial release and kinesio taping.
  Arms: CONTROL; MOPEXE
Other: MOPEXE — Transcutaneous Electrical Nerve Stimulation (TENS) treatment will be applied to the lumbar and suprapubic areas using 2 channels and 4 electrodes. Conventional TENS (120 Hz) will be applied simultaneously to the lumbar and suprapubic areas for 30 minutes. Hot pack application will be done sequentially to the lumbar and suprapubic areas for 15 minutes each, for a total of 30 minutes. 5 minute-Meditation Therapy 10 minute-Progressive Relaxation training ( Bernstein-Borkovec Method) 5 min - Breathing Exercises (Diaphragmatic Breathing Exercise, Pursed lip breathing Exercise) 35 min -Motor Imagery Technique Focused Pelvic Floor Exercises-MOPEXE 5 min - Meditation Therapy Twice a week for 60 minutes 12 weeks Participants will be evaluated online at the beginning of the research and at the end of the 12-week program.
  Arms: CONTROL; FEMOB
Other: CONTROL — Transcutaneous Electrical Nerve Stimulation (TENS) treatment will be applied to the lumbar and suprapubic areas using 2 channels and 4 electrodes. Conventional TENS (120 Hz) will be applied simultaneously to the lumbar and suprapubic areas for 30 minutes. Hot pack application will be done sequentially to the lumbar and suprapubic areas for 15 minutes each, for a total of 30 minutes.
  Arms: FEMOB; MOPEXE

SUMMARY:
42 women diagnosed with primary dysmenorrhea were included in the study and divided into three groups. the first group received treatment with a mobilization approach, the second group received motor imagery-focused exercises and the third group, as a control group received electrotherapy. all three groups received electrotherapy.

ELIGIBILITY:
Inclusion Criteria:

* primary dysmenorrhea

Exclusion Criteria:

* a contraindicated condition

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women
Enrollment: 42 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-02-03 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
McGill pain scale short form | 5 minutes
  The characteristic of pain felt by the patients during menstruation was evaluated using the McGill Pain Questionnaire-Short Form,With the McGill Melzack Pain Questionnaire, the location of the pain, the feeling it creates in the individual, its relationship with time, its severity and the level of viable pain for the individual are determined. High score indicates high level of pain

SECONDARY OUTCOMES:
Menstrual Attitude Questionnaire | 5 minutes
  The Turkish version of the Menstrual Attitude Scale (MBI) will be applied to determine the attitudes and behaviors of the participants during the menstrual period. Menstruation attitude scale includes 5 subtitles. These subheadings are;
  1. Menstruation as a debilitating event
  2. Menstruation as a bothersome event
  3. Menstruation as a natural event
  4. Ancipitation and prediction of the onset of menstruation
  5. Denial of any effect of menstruation
Functional and Emotional Dysmenorrhea Scale | 5 minutes
  This is a 14-item, 5-point Likert-type scale used to measure dysmenorrhea functionally and emotionally. There are no reverse items in the scale. The scale was developed to provide functional and emotional measurement of dysmenorrhea. As the scores obtained from the scale increase, the extent to which patients are functionally and emotionally affected by dysmenorrhea also increases.
Menstrual Symptom Questionnaire | 5 minutes
  The scale consists of 22 items that inquire about menstrual symptoms and is scored on a five-point Likert scale, from never (1) to always (5). The scale, which consists of three sub-dimensions, is evaluated in the sub-dimension of 'Negative effects/somatic complaints' with items 1-13, the sub-dimension of 'Menstrual pain symptoms' with items 14-19, and the sub-dimension of 'Coping methods' with items 20-22. An increase in the mean score indicates an increase in the severity of menstrual symptoms related to the relevant sub-dimension.
The Menstrual Distress Questionnaire | 5 minutes
  This is a self-reported assessment tool designed to comprehensively evaluate the physical and emotional symptoms experienced by individuals during their menstrual period. The scale consists of 25 questions, each with 5 sub-items, covering common symptoms such as abdominal pain, headache, nausea, irritability, and mood swings. Each item is scored using a Likert-type rating system to determine the frequency or severity with which the participant experiences the relevant symptom. As the total score on the scale increases, the intensity of the symptoms experienced during menstruation and their negative impact on daily life also increase. In this context, high scores indicate increased symptom severity and decreased quality of life. The scale offers a holistic assessment by encompassing both the somatic and emotional dimensions of menstruation-related symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Result] Toprak Celenay S, Kavalci B, Karakus A, Alkan A. Effects of kinesio tape application on pain, anxiety, and menstrual complaints in women with primary dysmenorrhea: A randomized sham-controlled trial. Complement Ther Clin Pract. 2020 May;39:101148. doi: 10.1016/j.ctcp.2020.101148. Epub 2020 Mar 18. PMID 32379680
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35419791/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37632569/